CLINICAL TRIAL: NCT07270354
Title: STUMBL (Study of the Management of Blunt Chest Wall Trauma) vs TTSS (Thoracic Trauma Severity Score) in Prediction of Morbidity and Mortality Rate of Blunt Chest Trauma
Brief Title: STUMBL vs TTSS in Predicting Morbidity and Mortality of Blunt Chest Trauma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Emad Ahmed Swefy, Emergency medicine resident at Assiut University, Assiut University
Other Study IDs: STUMBL-TTSS-BluntChestTrauma
Record Dates: First submitted 2025-11-20; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Blunt Chest Wall Trauma
Keywords: Blunt; Chest wall trauma; Emergency department
MeSH Terms: conditions — Emergencies | interventions — Diagnostic Imaging; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blunt Chest Trauma group: The Blunt Chest Trauma Cohort comprises all consecutive adult patients (≥18 years) presenting with blunt chest trauma to the Emergency Department of Assiut university between October 2025 and October 2026. Patients meeting inclusion criteria will be enrolled prospectively and followed throughout their hospital stay to record clinical course and outcomes. At presentation both the STUMBL and TTSS scores will be calculated for each patient using standard definitions. The cohort will be analyzed as a single group to evaluate the predictive performance of each score for predefined outcomes (morbidity and mortality)
  Interventions: Diagnostic Test: Chest X-Ray; Diagnostic Test: Computed Tomography (CT) Chest (with or without contrast)

INTERVENTIONS:
Diagnostic Test: Chest X-Ray — First-line imaging for suspected rib fractures, hemothorax, pneumothorax, or pulmonary contusion
Diagnostic Test: Computed Tomography (CT) Chest (with or without contrast) — Gold standard for detecting:
  Rib fractures (especially multiple and posterior).
  Pulmonary contusions and lacerations.
  Hemothorax, pneumothorax, hemopericardium.
  Pleural or mediastinal injuries

SUMMARY:
This study aim to compare the effectiveness of the STUMBL Score and the Thoracic Trauma Severity Score (TTSS) in predicting morbidity and mortality in patients with blunt chest wall trauma, and to evaluate which scoring system provides greater clinical utility for early risk stratification and management decisions.

DETAILED DESCRIPTION:
Blunt chest wall trauma poses a clinical challenge due to its substantial contribution to morbidity and mortality, particularly following falls and vehicular accidents. Early identification of patients at high risk of complications is critical yet difficult, as delayed respiratory issues often escape initial detection. Traditional trauma scoring systems (e.g. ISS, AIS) lack specificity for isolated thoracic injury, creating a niche for more focused prognostic tools.

Two promising models have emerged: the STUMBL Score-based on age, number of rib fractures, chronic lung disease, pre-injury anticoagulant use, and oxygen saturation-is explicitly designed for blunt chest trauma prognosis. Studies report strong discriminatory performance, with development-phase c-index up to 0.96 . External validations vary: one UK cohort showed STUMBL ≥ 11 had a sensitivity of 79%, specificity of 78%, and AUC of 0.84-comparable to clinician judgment ; Italian data demonstrated excellent discrimination (C-index ~0.90) and calibration .

The Thoracic Trauma Severity Score (TTSS), initially validated in polytrauma ICU patients, yields moderate to good discrimination (c-indices 0.72-0.85) across validation studies .

Though these scores show promise, high methodological bias and limited external validations temper their widespread adoption . A direct, comparative analysis of STUMBL and TTSS within a well-defined patient cohort is thus needed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) presenting with blunt chest trauma.
* Patients who have given written informed consent to participate in the study

Exclusion Criteria:

* Penetrating chest injuries
* Pediatric patients (<18 years)
* Patients with incomplete records or who decline consent
* Pregnant women
* Disturbed conscious patients
* Mechanically ventilated patients
* Polytrauma patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients presenting with blunt chest trauma to the Emergency Department of Assiut university during the study period from October 2025 to October 2026
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
To compare the predictive accuracy of the STUMBL score and TTSS in forecasting morbidity and mortality in patients with blunt chest trauma | 14 day duration follow-up after ED admission

SECONDARY OUTCOMES:
Easy of use of STUMBL score and TTSS score in emergency clinical settings | 14 day duration follow-up after ED admission
  How measured:
  Completion time measured with a stopwatch (minutes)
To correlate each score with specific outcomes such as pneumonia, need for mechanical ventilation, ICU admission, and in-hospital mortality | 14 day duration follow-up after ED admission

CONTACTS AND LOCATIONS:
Overall Officials: Jehan Ahmed Sayed, Professor of Anathesia and ICU, Principal Investigator — Assiut University; Yasmin Elsayed Mohamed Elbeltagy, Lecturer of emergency medicine, Study Director — Seuz canal University

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is conducted as part of an academic thesis project. Data are limited to internal use within the research team and protected by institutional and ethical regulations

REFERENCES:
- [Result] Seok J, Cho HM, Kim HH, Kim JH, Huh U, Kim HB, Leem JH, Wang IJ. Chest Trauma Scoring Systems for Predicting Respiratory Complications in Isolated Rib Fracture. J Surg Res. 2019 Dec;244:84-90. doi: 10.1016/j.jss.2019.06.009. Epub 2019 Jul 4. PMID 31279998
- [Result] Baddam S, Burns B. Systemic Inflammatory Response Syndrome. 2025 Jun 20. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK547669/ PMID 31613449
- [Result] Callisto E, Costantino G, Tabner A, Kerslake D, Reed MJ. The clinical effectiveness of the STUMBL score for the management of ED patients with blunt chest trauma compared to clinical evaluation alone. Intern Emerg Med. 2022 Sep;17(6):1785-1793. doi: 10.1007/s11739-022-03001-0. Epub 2022 Jun 23. PMID 35739456